CLINICAL TRIAL: NCT01625286
Title: A Phase I/II Study of AZD5363 Combined With Paclitaxel in Patients With Advanced or Metastatic Breast Cancer. Comprising a Safety Run-In and a Placebo-controlled Randomised Expansion in ER+ve Patients Stratified by PIK3CA Mutation Status
Brief Title: Investigating Safety, Tolerability and Efficacy of AZD5363 When Combined With Paclitaxel in Breast Cancer Patients
Acronym: BEECH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3610C00002; 2011-006312-31 (EudraCT Number)
Record Dates: First submitted 2012-05-10; First posted 2012-06-21 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Advanced or Metastatic Breast Cancer; ER+ve Advanced or Metastatic Breast Cancer
Keywords: advanced breast cancer,; metastatic breast cancer,; ER+ve breast cancer,; Estrogen receptor positive breast cancer,; PIK3CA mutated advanced or metastatic breast cancer; AKT inhibitor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A: Intermittent schedule (2/5) (Experimental): See intervention description below.
  Interventions: Drug: AZD5363 when combined with weekly paclitaxel.
- Part A: Intermittent schedule (4/3) (Experimental): See intervention description below.
  Interventions: Drug: AZD5363 when combined with weekly paclitaxel.
- Part B: AZD5363 combined with paclitaxel (Active Comparator): See intervention description below.
  Interventions: Drug: AZD5363when combined with weekly paclitaxel.
- Part B: paclitaxel combined with placebo (Placebo Comparator): See intervention description below.
  Interventions: Drug: A placebo in combination with weekly paclitaxel.

INTERVENTIONS:
Drug: AZD5363 when combined with weekly paclitaxel. — AZD5363: oral capsule, twice daily in a weekly 2 days on-treatment, 5 days-off, schedule. Treatment to begin the day following the first dose of paclitaxel and to continue until treatment withdrawal. Paclitaxel: intravenously once a week. AZD5363 and paclitaxel will be received for 3 consecutive weeks, followed by one week off-therapy in 4-week cycles.
  Arms: Part A: Intermittent schedule (2/5)
Drug: AZD5363 when combined with weekly paclitaxel. — AZD5363: oral capsule, twice daily in a weekly 4 days on-treatment, 3 days-off, schedule. Treatment to begin the day following the first dose of paclitaxel and to continue until treatment withdrawal. Paclitaxel: intravenously once a week. AZD5363 and paclitaxel will be received for 3 consecutive weeks, followed by one week off-therapy in 4-week cycles.
  Arms: Part A: Intermittent schedule (4/3)
Drug: AZD5363when combined with weekly paclitaxel. — Either a 2/5 or 3/4 intermittent dosing schedule of AZD5363 based on the outcome of Part A. Dosage: oral formulation, twice daily. Treatment to begin the day following the first dose of paclitaxel and to continue until treatment withdrawal. Paclitaxel: intravenously once a week. AZD5363 and paclitaxel will be received for 3 consecutive weeks, followed by one week off-therapy in 4-week cycles.
  Arms: Part B: AZD5363 combined with paclitaxel
Drug: A placebo in combination with weekly paclitaxel. — Either a 2/5 or 3/4 intermittent dosing schedule of placebo matched to AZD5363 based on the outcome of Part A. Dosage: oral formulation, twice daily. Treatment to begin the day following the first dose of paclitaxel and to continue until treatment withdrawal. Paclitaxel: intravenously once a week. placebo and paclitaxel will be received for 3 consecutive weeks, followed by one week off-therapy in 4-week cycles.
  Arms: Part B: paclitaxel combined with placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of different doses and schedules of AZD5363, when in combination with paclitaxel, in treatment of patients with advanced or metastatic breast cancer. Also to investigate a selected dose and schedule of AZD5363 in combination with paclitaxel vs. paclitaxel in combination with placebo in treatment of patients with estrogen receptor-positive advanced or metastatic breast cancer, including a subgroup who have the phosphoinositide-3-kinase, catalytic, alpha polypeptide (PIK3CA) tumour mutation.

DETAILED DESCRIPTION:
This is a Phase I/II multicentre, study investigating the safety, tolerability and efficacy of a twice-daily oral formulation of AZD5363 when combined with a weekly intravenous paclitaxel infusion in patients with advanced or metastatic breast cancer. Study treatment is given in 28-day cycles, comprising three weeks on-therapy followed by one week off-therapy.

The study will be conducted in two parts:

Part A. Approximately 40 patients will be recruited to this Phase I multiple ascending-dose safety run-in evaluation of each of two intermittent dosing schedules (2 days per week or 4 days per week) of AZD5363 given in combination with weekly paclitaxel. The study population is female patients, 18 years or older, with advanced or metastatic breast cancer.

The purpose of Part A is to assess the comparative safety, tolerability, pharmacokinetics and preliminary efficacy of both schedules to determine one dose and schedule of AZD5363 to take forward to study Part B in combination with weekly paclitaxel.

Part A assessments will be made in dose-escalating cohorts of 3 to 6 patients to determine a recommended dose in each of the schedules. A total of 6 patients must be evaluated at a selected dose level for it to be confirmed as the recommended dose. All dose evaluations and recommendations will be conducted by a Safety Review Committee.

Part A Patients will undergo assessments up to to withdrawal from the study or to discontinuation of study therapy.

Part B. A minimum of 100 patients will be recruited to this Phase II double-blind, placebo-controlled, stratified and randomised evaluation of two treatment regimens: AZD5363 (at a dose selected and schedule from Part A) in combination with weekly paclitaxel vs. weekly paclitaxel plus placebo. The study population is female patients with Estrogen Receptor Positive advanced or metastatic breast cancer; of which approximately 50 will have the phosphoinositide-3-kinase, catalytic, alpha polypeptide (PIK3CA) mutation.

Part B patients will be stratified by PIK3CA tumour mutation status as: tumour mutation positive or tumour mutation not-detected. Under each stratum patients will be randomised to receive either paclitaxel + AZD5363 or paclitaxel + placebo.

The purpose of Part B is to assess relative efficacy of both active and placebo regimens by comparison of: progression-free survival, overall survival, tumour response, safety and tolerability in the overall ER+ve advanced or metastatic breast cancer population, and in a subgroup of these patients with the PIK3CA tumour mutation. Patient safety and therapy tolerability will be monitored by an independent Safety Review Committee throuighout the course of Part B.

Part B patients will be followed for assessment of overall survival, or to withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Female patient.
* Aged at least 18 years.
* Histological or cytological confirmation of breast cancer with evidence of advanced or metastatic disease (must be ER+ve, HER2-ve, in Part B).
* World Health Organisation (WHO) performance status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks.

Exclusion Criteria:

* Clinically significant abnormalities of glucose metabolism.
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable (not requiring steroids).
* Evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses or active infections including hepatitis B, C and HIV.
* Any prior exposure to agents which inhibit AKT as the primary pharmacological activity.
* Part A: more than two prior courses of chemotherapy (including taxanes) for advanced or metastatic breast cancer.

Part B: any prior chemotherapy for advanced or metastatic breast cancer.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-10-03 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lindemann, MBChB MBA, Study Director — AstraZeneca
Locations (35):
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Research Site, Brno, Czechia
- France (3):
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Villejuif
- Japan (6):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Mitaka-shi
  - Research Site, Osaka
  - Research Site, Ōita
- Mexico (4):
  - Research Site, Estado de México
  - Research Site, Juchitán
  - Research Site, Monterrey
  - Research Site, Oaxaca City
- Peru (2):
  - Research Site, Lima
  - Research Site, Miraflores
- Research Site, Singapore, Singapore
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Valencia
- United Kingdom (6):
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Plymouth
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Hrebien S, Citi V, Garcia-Murillas I, Cutts R, Fenwick K, Kozarewa I, McEwen R, Ratnayake J, Maudsley R, Carr TH, de Bruin EC, Schiavon G, Oliveira M, Turner N. Early ctDNA dynamics as a surrogate for progression-free survival in advanced breast cancer in the BEECH trial. Ann Oncol. 2019 Jun 1;30(6):945-952. doi: 10.1093/annonc/mdz085. PMID 30860573
- [Derived] Turner NC, Alarcon E, Armstrong AC, Philco M, Lopez Chuken YA, Sablin MP, Tamura K, Gomez Villanueva A, Perez-Fidalgo JA, Cheung SYA, Corcoran C, Cullberg M, Davies BR, de Bruin EC, Foxley A, Lindemann JPO, Maudsley R, Moschetta M, Outhwaite E, Pass M, Rugman P, Schiavon G, Oliveira M. BEECH: a dose-finding run-in followed by a randomised phase II study assessing the efficacy of AKT inhibitor capivasertib (AZD5363) combined with paclitaxel in patients with estrogen receptor-positive advanced or metastatic breast cancer, and in a PIK3CA mutant sub-population. Ann Oncol. 2019 May 1;30(5):774-780. doi: 10.1093/annonc/mdz086. PMID 30860570
- See also: CSPandAmendments_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1362&filename=CSPandAmendments_redacted.pdf
- See also: SAP_PartAandB_redactedsignature — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1362&filename=SAP_PartAandB_redactedsignature.pdf
- See also: SAP_PartAandB_redactedsignature — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1362&filename=SAP.pdf
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3610C00002&attachmentIdentifier=6c54545e-f7c7-4077-b74d-f33da44c4436&fileName=D3610C00002_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Schedule 1 560 mg bd: Schedule 1 - AZD5363 560 mg bd (2 days on/5 days off) with Paclitaxel 90 mg/m2 once weekly. 3/4 weeks.
- Part A Schedule 1 640 mg bd: Schedule 1 - AZD5363 640 mg bd (2 days on/5 days off) with Paclitaxel 90 mg/m2 once weekly. 3/4 weeks.
- Part A Schedule 2 360 mg bd: Schedule 2 - AZD5363 360 mg bd (4 days on/3 days off) with Paclitaxel 90 mg/m2 once weekly. 3/4 weeks.
- Part A Schedule 2 400 mg bd: Schedule 2 - AZD5363 400 mg bd (4 days on/3 days off) with Paclitaxel 90 mg/m2 once weekly. 3/4 weeks.
- Part A Schedule 2 480 mg bd: Schedule 2 - AZD5363 480 mg bd (4 days on/3 days off) with Paclitaxel 90 mg/m2 once weekly. 3/4 weeks.
- Part B AZD5363; Part B Placebo: (4 days on/3 days off) with Paclitaxel 90 mg/m2 once weekly
Period: Overall Study
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Started (RANDOMIZATION CODE ALLOCATED) | 12 | 8 | 5 | 7 | 6 | 54 | 56
Received AZD5363/Placebo Treatment | 12 | 8 | 5 | 7 | 6 | 54 | 55
Did Not Receive AZD5363/Placebo Trt | 0 | 0 | 0 | 0 | 0 | 0 | 1
Completed (Completed Study includes patients who were on study or treatment at the final database lock for primary analysis) | 6 | 4 | 0 | 0 | 0 | 40 | 37
Not Completed | 6 | 4 | 5 | 7 | 6 | 14 | 19
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 11 | 16
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Any reason not specifically recorded | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive disease | 6 | 3 | 4 | 5 | 5 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients with data who were included in the full analysis set for Part A and the intention to treat analysis set in Part B'
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo | Total
Number analyzed (Participants) | 12 | 8 | 5 | 7 | 6 | 54 | 56 | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (9.92) | 58.8 (12.78) | 56.6 (10.26) | 47.1 (9.41) | 49.8 (13.12) | 54.3 (10.01) | 57.4 (11.38) | 58.8 (11.24)
Age, Customized [Count of Participants; unit: Participants] — Population: For Part A Schedule 2 400 mg bd, there were no participants aged >=65
  Participants
    <50 | 5 | 3 | 1 | 4 | 2 | 19 | 16 | 50
    >=50 - <65 | 5 | 2 | 3 | 3 | 3 | 24 | 26 | 66
    >=65 | 2 | 3 | 1 | 0 | 1 | 11 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 5 | 7 | 6 | 54 | 56 | 148
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 0 | 12 | 15 | 28
  Black Or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 10 | 8 | 5 | 7 | 6 | 24 | 18 | 78
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 15 | 16 | 31
  Other | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity (DLT) Events - Part A
Description: An Adverse Event (AE) or laboratory abnormality considered to be related to study drug, that starts at any time during the DLT evaluation period (Cycle 1) and is dose limiting
Time Frame: During Part A DLT evaluation period (Cycle 1, up to 28 days)
Population: All Part A patients who either completed the DLT evaluation period with at least 80% of specified dose (of AZD5363 or paxlitaxel) or who experienced a DLT. DLT events were not assessed for Part B participants.
Measure: Number; unit: participants
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 11 | 6 | 5 | 7 | 6 | 0 | 0
participants | 0 | 2 | 0 | 0 | 2 |  |

2. Primary Outcome: Progression Free Survival (PFS) - Part B
Description: Time from randomisation to date of objective disease progression or death (by any cause in the absence of progression). Progression defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a >= 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on the study, and an absolute increase of >=5mm, or progression of non-target lesions or the appearance of new lesions.
Time Frame: From randomisation date to date of objective disease progression or death (by any cause) whichever came first, assessed every 12 wks (median total treatment duration AZD5363=325.5 days; Placebo=245 days)
Population: Intent to Treat (ITT), all randomised patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 54 | 56
Months |  |  |  |  |  | 10.9 [8.3 to 12.4] | 8.4 [8.2 to 10.8]
Statistical Analysis 1: Comparison: Part B AZD5363 vs Part B Placebo; Test type: Superiority — A hazard ratio < 1 favours AZD5363; p = 0.308, Regression, Cox — 2-sided p-value; Cox PH model including treatment and PIK3CA status as factors/covariates; Hazard Ratio (HR) = 0.80, 80% CI 2-sided [0.60 to 1.06]

3. Secondary Outcome: Change in Tumour Size at 12 Weeks
Description: Percentage change from baseline to week 12 in sum of longest diameters of target lesions as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1). Based on patients with measurable disease who had sufficient data available to either calculate or impute a change at 12 weeks
Time Frame: RECIST tumour assessments every 12 weeks
Population: Part A:Full Analysis Set (FAS) Part B: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 10 | 7 | 5 | 5 | 4 | 53 | 55
% change from baseline | -11.0 (33.42) | -15.7 (13.33) | -19.1 (17.73) | -18.3 (37.74) | -10.2 (24.84) | -34.2 (28.91) | -25.4 (35.87)
Statistical Analysis 1: Comparison: Part B AZD5363 vs Part B Placebo; Test type: Superiority; p = 0.081, ANCOVA — 1-sided p-value; Mean Difference (Final Values) = -8.9, 80% CI 2-sided [-17.1 to -0.8]

4. Secondary Outcome: Objective Response Rate (ORR) at Week 12
Description: Percentage of patients who have at least one visit response of Complete Response or Partial Response prior to any evidence of progression at week 12 as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) for target lesions (TL) and assessed by MRI or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Complete Response (CR), disappearance of all target lesions, any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm; Objective Response Rate (ORR) = CR + PR
Time Frame: RECIST tumour assessments every 12 weeks
Population: Part A:Full Analysis Set (FAS) Part B: Intent to Treat (ITT)
Measure: Number; unit: % of participants
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 12 | 8 | 5 | 7 | 6 | 54 | 56
% of participants | 41.7 | 12.5 | 0 | 0 | 0 | 50 | 42.9

5. Secondary Outcome: Best Objective Response (BOR)
Description: Number of patients, taking their BOR, which is their best objective tumour response based on RECIST measurements throughout the whole study as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) for target lesions (TL) and assessed by MRI or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Complete Response (CR), disappearance of all target lesions, any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm.
Time Frame: From date of randomisation, assessed every 12 weeks (median total treatment duration AZD5363 = 325.5 days; Placebo = 245 days).
Measure: Number; unit: Participants
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 12 | 8 | 5 | 7 | 6 | 54 | 56
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 3 | 4
  Partial Response (PR) | 0 | 2 | 1 | 1 | 0 | 29 | 28
  Stable Disease (SD) | 7 | 4 | 3 | 4 | 3 | 14 | 14
  Progression | 4 | 1 | 1 | 1 | 2 | 6 | 8
  Not Evaluable (NE) | 1 | 1 | 0 | 1 | 1 | 2 | 2

6. Secondary Outcome: Overall Objective Response Rate
Description: Percentage of patients, taking their best objective tumour response based on RECIST measurements throughout the whole study as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) for target lesions (TL) and assessed by MRI or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Complete Response (CR), disappearance of all target lesions, any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm. Overall Response Rate (ORR) = CR + PR
Time Frame: as for outcome 5
Population: Part A:Full Analysis Set (FAS) Part B: Intent to Treat (ITT)
Measure: Number; unit: % of participants
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 12 | 8 | 5 | 7 | 6 | 54 | 56
% of participants | 0 | 25 | 20 | 14.3 | 0 | 59.3 | 57.1

7. Secondary Outcome: Number of Subjects Without Progression Disease at Week 12 - Part A
Description: Percentage of patients with a 12 week visit response of CR, PR or SD (as defined by RECIST 1.1) with no evidence of previous progression as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) for target lesions (TL) and assessed by MRI or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Complete Response (CR), disappearance of all target lesions, any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm.
Time Frame: up to 12 weeks
Population: Part A Full Analysis Set (FAS). Not recorded in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 12 | 8 | 5 | 7 | 6 | 0 | 0
Participants | 6 | 5 | 3 | 4 | 2 |  |

8. Secondary Outcome: Duration of Response (DOR) - Part B
Description: Date of first documentation of response (Complete Response/Partial Response) until the date of disease progression as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) for target lesions (TL) and assessed by MRI or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Complete Response (CR), disappearance of all target lesions, any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm.. If a subject does not progress following a response, then their DOR will use the PFS censoring time.
Time Frame: as for outcome 5
Population: Part B, all patients with a response in the ITT analysis set. Not collected in Part A
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 54 | 56
Months |  |  |  |  |  | 8.3 [6 to 11.3] | 8.2 [5.6 to 10.6]

9. Secondary Outcome: Durable Response Rate (DRR) - Part B
Description: Percentage of patients who have a Complete Response (CR) or Partial Response (PR) lasting continuously for at least 24 weeks as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) for target lesions (TL) and assessed by MRI or CT: PR, >=30% decrease in the sum of the longest diameter of target lesions; CR, disappearance of all target lesions, any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm.
Time Frame: as for outcome 5
Population: Part B, ITT analysis set. Not collected in Part A
Measure: Number; unit: % of participants
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 54 | 56
% of participants |  |  |  |  |  | 48.1 | 37.5
Statistical Analysis 1: Comparison: Part B AZD5363 vs Part B Placebo; Test type: Superiority; p = 0.139, Regression, Logistic — 1-sided p-value; including treatment and PIK3CA status as factors/covariates; Odds Ratio (OR) = 1.53, 80% CI 2-sided [0.93 to 2.54]

10. Secondary Outcome: Overall Survival - Part B
Description: The interval between the date of randomisation and the date of patient death due to any cause. All Part B patients were analysed, number of deaths is presented.
Time Frame: From date of randomisation, assessed every 12 weeks, up until the time of final statistical analysis. (median total treatment duration AZD5363 = 325.5 days; Placebo = 245 days).
Population: Part B Intent to Treat (ITT). Not collected in Part A
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A Schedule 1 560 mg bd | Part A Schedule 1 640 mg bd | Part A Schedule 2 360 mg bd | Part A Schedule 2 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 54 | 56
months |  |  |  |  |  | 32.8 [21.3 to 32.8] | NA [20.9 to NA] — NA = The median OS and the upper 95% Confidence limit were both non calculable
Statistical Analysis 1: Comparison: Part B AZD5363 vs Part B Placebo; Test type: Superiority — A hazard ratio < 1 favours AZD5363; p = 0.482, Log Rank — 2-sided p-value; Cox PH model including treatment and PIK3CA status as factors/covariates; Hazard Ratio (HR) = 0.77, 80% CI 2-sided [0.48 to 1.24]

ADVERSE EVENTS:
Time Frame: Time of signature of informed consent throughout the treatment period up to and including the follow-up period (median follow-up AZD5363 16.9 months; Placebo 15.2 months)
Description: The 5% threshold is applied to treatment schedule in Part A and then the Part A AEs are labelled as MedDRA v20.0 (schedule 1) or MedDRA v18.1 (schedule 2). The 5% threshold is applied to each Part B treatment arm and then the Part B AEs are labelled as MedDRA v19.1 One patient in the placebo group did not receive placebo treatment (hence n=56 for All Cause Mortality but n=55 for SAEs and Other AEs)
Groups:
- Sched 1 - AZD5363 640 mg bd: (2 days on/5 days off) with Paclitaxel 90 mg/m2 once weekly. 3/4 weeks.
- Sched 2 - AZD5363 360 mg bd; Sched 2 - AZD5363 400 mg bd: (4 days on/3 days off) with Paclitaxel 90 mg/m2 once weekly. 3/4 weeks.
Arm/Group | Part A Schedule 1 560 mg bd | Sched 1 - AZD5363 640 mg bd | Sched 2 - AZD5363 360 mg bd | Sched 2 - AZD5363 400 mg bd | Part A Schedule 2 480 mg bd | Part B AZD5363 | Part B Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8 | 1/5 | 1/7 | 0/6 | 13/54 | 15/56
Serious Adverse Events (participants affected / at risk) | 3/12 | 3/8 | 0/5 | 1/7 | 4/6 | 13/54 | 8/55
Other Adverse Events (participants affected / at risk) | 12/12 | 8/8 | 5/5 | 7/7 | 6/6 | 50/54 | 48/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Schedule 1 560 mg bd (N=12) | Sched 1 - AZD5363 640 mg bd (N=8) | Sched 2 - AZD5363 360 mg bd (N=5) | Sched 2 - AZD5363 400 mg bd (N=7) | Part A Schedule 2 480 mg bd (N=6) | Part B AZD5363 (N=54) | Part B Placebo (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Schedule 1 560 mg bd (N=12) | Sched 1 - AZD5363 640 mg bd (N=8) | Sched 2 - AZD5363 360 mg bd (N=5) | Sched 2 - AZD5363 400 mg bd (N=7) | Part A Schedule 2 480 mg bd (N=6) | Part B AZD5363 (N=54) | Part B Placebo (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (31) | 6 (34) | 6 (101) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (8) | 2 (5) | 5 (15) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 4 (9) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (4) | 6 (11) | 3 (3) | 0 (0) | 0 (0)
Device breakage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (6) | 0 (0) | 2 (3) | 2 (5) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (32) | 15 (20)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (16) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (21) | 7 (26)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 41 (228) | 15 (32)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 8 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 21 (33) | 13 (19)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (26) | 4 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (20) | 8 (10)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 7 (16)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (20) | 11 (14)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (8)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 8 (11)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (15) | 3 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (11) | 5 (7)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 3 (3)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (13) | 5 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 5 (6)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 13 (22) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 11 (19) | 4 (6)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 4 (8) | 3 (5)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (18)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (48) | 6 (13)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 5 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 12 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (13) | 7 (8)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (14) | 10 (12)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 13 (22) | 18 (26)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (17) | 10 (11)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (13) | 8 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 9 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 6 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 28 (28) | 27 (30)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 4 (4)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (7)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 4 (8)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (18) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (10)
Anaemia (Blood and lymphatic system disorders) | 6 (17) | 4 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (20) | 3 (23) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 11 (66) | 7 (57) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 2 (5) | 0 (0) | 2 (2) | 3 (10) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (17) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 6 (12) | 5 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroxine decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (39) | 3 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 5 (7) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (13) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (6) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Melanoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (23) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear canal erythema (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival pallor (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver palpable (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calcium deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
QoL, PK/PD & efficacy response modelling were considered non-key secondary endpoints and not disclosed at this time. QoL data was limited and considered exploratory, PK/PD and modelling were not reported in CSR. Diarrhoea burden is reported with AEs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-02-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT01625286/Prot_002.pdf
  • Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT01625286/SAP_001.pdf